CLINICAL TRIAL: NCT03863158
Title: Optimal Timing of Coronary Artery Bypass Grafting in Hemodynamically Stable Patient After Myocardial Infarction and Definition of Poor Prognostic Factors. Pilot Study
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier La Chartreuse (Other)
Collaborators: BOUCHOT Olivier (Unknown); LAUBRIET-JAZAYERI Aline (Unknown)
Responsible Party: Principal Investigator, MORGANT Marie-Catherine, Principal investigator, Centre Hospitalier La Chartreuse
Other Study IDs: CCVT-ChloéBernard 2019
Record Dates: First submitted 2019-03-01; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Cardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention / medical records only

SUMMARY:
Acute coronary syndromes (ACS) represent the leading cause of death in France. Their incidence is increasing due to population aging and to the persistence of cardiovascular risk factors. Currently, revascularization surgery remains outside the emergency treatment, because early performed, it tends to lead to extension and hemorrhage of the infarcted area, because of the CPB, aortic clamping, cardioplegia, and other heart manipulation.

However, CABG are indicated as an emergency in some situations of STEMI: Threat of infarction of an extended territory without favorable anatomy to angioplasty, anatomy not favorable to angioplasty associated with cardiogenic shock or persistent ischemia, acute complications of myocardial infarction (massive mitral insufficiency, interventricular communication, parietal rupture) requiring surgery under CPB with concomitant bypass surgery or failure of angioplasty (proximal coronary dissection).

Operative mortality is high; 15 to 20% for patients operated 12 to 48 hours after AMI and 4-5% for those operated after 48 hours.

Nevertheless, it seems legitimate to study if there would be a place for primary surgical revascularization in case of patient with hemodynamically stable ACS, in order to limit myocardial ischemia, spread of necrosis, to limit the risk of recurrence, and the consequences of low cardiac output. Performing a complete early surgical revascularization could limit the ischemia-reperfusion syndrome and anticipate the occurrence of cardiogenic shock.

DETAILED DESCRIPTION:
Trial on medical records only

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting acute myocardial infarction with hemodynamic stability at the diagnosis
* Patients undergoing coronary artery bypass in Dijon University hospital

Exclusion Criteria:

* Patients with Acute pulmonary oedema
* Patients with cardiorespiratory arrest before coronary angiography
* hemodynamically unstable patient at diagnosis
* patients requiring combined surgery
* patients with unstable angina

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective Observationnal study (medical records only) on patients undergoing CABG in emergency from the 2007 January 1 to 2018 december 31.
Sampling Method: Non-Probability Sample
Enrollment: 476 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Correlation between the mortality rate and the delay between the surgical revascularization and the date of diagnosis of mycardial infaction in hemodynamically stable patients | 30 days
  Delay in days between diagnosis and surgery

SECONDARY OUTCOMES:
Determine the predictors of intra-hospital mortality rate in hemodynamically stable patients operated of coronary bypass | 30 days
  Evaluate the results of evaluations carried out in patients who died compared to patients who did not die and the normal population

IPD SHARING:
Plan to Share IPD: No
Screening of patients will be done from lists of patients who have undergone emergency coronary bypass surgery Demographic, clinical, paraclinical and biological data of patients will be collected internally using the data available in the computerized patient record of Dijon University Hospital (DxCare).
  The data will be collected in an Excel file, which is hosted by the CHU server. As this is a monocentric observational study, it is not envisaged that the data will be transferred outside Dijon University Hospital.